CLINICAL TRIAL: NCT03248674
Title: Diagnostic Performance of Coronary Computed Tomography Angiography With Computed Tomography Fractional Flow Reserve in Kidney Transplantation Candidates
Brief Title: Diagnostic Performance of Coronary CT Angiography With CT FFR in Kidney Transplantation Candidates
Status: Terminated | Type: Observational
Why Stopped: Difficulty with recruitment in this patient population.
Sponsor: Stanford University (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Dominik Fleischmann, MD, Professor of Radiology, Stanford University
Other Study IDs: IRB-41455
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Disease; Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: CT FFR — CT FFR calculated the fractional flow reserve based on the data derived for a regular coronary CT angiography. Computation is based on development of an anatomic model of the epicardial coronary arteries for each case and calculating the maximum coronary flow during maximal hyperaemia based on a mathematical model incorporating fluid dynamics. These post-processing steps require quantification of the patient-specific myocardial mass as this allows for an estimation of the baseline coronary blood flow.

SUMMARY:
Patients with chronic kidney disease (CKD) before kidney transplantation require that obstructive coronary artery disease (CAD) is excluded, as cardiovascular complications are the leading cause of mortality in kidney transplant patients. However, in this patient population, the optimal method for the detection of obstructive CAD has not been identified. Noninvasive stress tests such as Dobutamine stress echocardiography or nuclear perfusion study have low diagnostic accuracy. CT fractional flow reserve measurement (CT FFR) is a novel non-invasive (FDA approved) imaging test to identify obstructive CAD. The goal of this project is to evaluate the diagnostic accuracy of CT FFR in the detection of obstructive coronary artery disease in patients with chronic kidney disease before kidney transplantation.

DETAILED DESCRIPTION:
Transplantation is the therapy of choice for most patients with stage 5 chronic kidney disease (CKD) and end stage renal disease (ESRD). Kidney transplantation improves quality of life and overall survival rates. Cardiovascular disease is the most common complication and leading cause of death in the transplant population. In order to assess the risk of cardiac events perioperatively and after kidney transplantation, the majority of kidney transplantation candidates undergo cardiac evaluation, including non-invasive cardiac stress imaging or invasive coronary angiography before transplantation. Invasive coronary angiography is associated with small but definite risk of bleeding or myocardial infarction, making non-invasive cardiac stress imaging such as dobutamine stress echocardiography (DSE) or nuclear myocardial perfusion scintigraphy (MPS) the preferred method. However, non-invasive cardiac stress imaging in patients with stage 5 CKD and ESRD demonstrates only moderate accuracy. DSE and MPS showed only sensitivities ranging from 0.44 to 0.89 and from 0.29 to 0.92, respectively, for identifying one or more severe coronary artery stenosis (defined as coronary diameter stenosis of more than 70%). Due to the moderate accuracy, several transplant centers (including Stanford) still continue to rely on invasive coronary angiography for their populations instead of non-invasive cardiac testing. Thus improved non-invasive cardiac testing with higher sensitivities and specificity are highly desirable in this patient population.

A promising alternative is the use of coronary CT angiography (cCTA) in combination with CT based fractional flow reserve (CT-FFR). Non-invasive cCTA alone has recently been evaluated in kidney transplantation candidates. It demonstrated high sensitivity (0.93) but limited specificity (0.63) in the detection of obstructive coronary artery disease, most likely related to the high prevalence of coronary artery calcifications in patients with CKD and ESRD. The specificity of coronary CTA can be improved by a new image analysis techniques, which allow the calculation of the hemodynamic significance - expressed as the relative pressure drop across a lesion similar - based on computational fluid dynamics derived from the conventional coronary CTA (6). In various study populations, the combination of coronary CT angiography and CT FFR showed excellent correlation with invasive FFR derived from invasive coronary angiography, which is the current gold standard. The implementation of CT- FFR has shown an improvement of the specificity of coronary CTA , even in the presence of coronary artery calcifications. However, no study so far assessed the diagnostic accuracy of coronary angiography with CT-FFR in candidates for kidney transplantation.

Goal The objective of this project is to evaluate and establish a new non-invasive cardiac test in the detection of coronary artery disease for candidates before kidney transplantation.

Specific Aims We want to confirm the promising results of CT FFR in this specific patient population and want to establish an alternative non-invasive cardiac test.

Study Design This study is designed as a prospective observational cohort study with a study population of 50 -100 patients. All patients who are included in this study will undergo coronary CT angiography with CT-FFR (research part) and a clinically indicated invasive coronary angiography with invasive FFR (standard of care). Coronary angiography and invasive FFR will act as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for kidney transplantation on dialysis without any residual kidney function AND referred to invasive coronary angiography for cardiac evaluation
* Referral to invasive coronary angiography is based on algorithm used at the Transplant Readiness Assessment Clinic (TRAC) at Stanford:
* A. Diabetic Candidates older than 45 years.
* B. Diabetic Candidates under 45 years old and any one of the following criteria is present:
* a) 25 year History of Diabetes
* b) 5 year Smoking History
* c) Abnormal EKG (ST-T wave changes)

Exclusion Criteria:

* Hemodynamically and clinically unstable condition (angina at rest, malignant arrhythmias)
* Known ischemic heart disease (prior, documented myocardial infarction, prior stenting or coronary artery bypass graft surgery)
* BMI>30 kg/m2, or weight >120 kg.
* Atrial fibrillation or other arrhythmia, >6 ectopic beats per minute
* Known or suspected allergy to iodinated contrast medium
* Pregnancy cannot be excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for kidney transplantation without any residual kidney function and referred to cardiac evaulation.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CT FFR. | CT FFR and Invasive FFR are calculated immediately after coronary CT angiography and invasive coronary angiography
  Diagnostic accuracy of CT FFR (per vessel) in the detection of hemodynamically significant CAD as compared to invasive FFR derived from invasive coronary angiography (reference standard). Presence or absence of hemodynamically significant coronary artery disease in concordance between CT FFR and invasive FFR. Hemodynamically significant stenosis is defined as CT FFR value below 0.8.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Fleischmann, M.D., Principal Investigator — Stanford Radiology
Locations (1):
- Stanford Healthcare, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No